CLINICAL TRIAL: NCT00646529
Title: A Six Month, Randomized, Open-Label, Safety Study of Symbicort (160/4.5mcg) Compared to Pulmicort Turbuhaler in Asthmatic Children Aged Six to Eleven Years - SAPLING
Brief Title: Long-Term Safety of Symbicort in Asthmatic Children - SAPLING
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SD-039-0719; D5896C00719
Record Dates: First submitted 2008-03-26; First posted 2008-03-28 (Estimated); Last update posted 2009-03-30 (Estimated); Status verified 2009-03

CONDITIONS: Asthma
Keywords: asthma; children; Symbicort; budesonide/formoterol; Pulmicort; budesonide
MeSH Terms: conditions — Asthma | interventions — Budesonide; Formoterol Fumarate; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): budesonide/formoterol
  Interventions: Drug: budesonide/formoterol (Symbicort)
- 2 (Active Comparator): budesonide
  Interventions: Drug: budesonide (Pulmicort)

INTERVENTIONS:
Drug: budesonide/formoterol (Symbicort)
  Other Names: Symbicort
  Arms: 1
Drug: budesonide (Pulmicort)
  Other Names: Pulmicort
  Arms: 2

SUMMARY:
The purpose of this study is to assess the safety of Symbicort compared to Pulmicort in asthmatic children aged 6 to 11 years

ELIGIBILITY:
Inclusion Criteria:

* At least 6 and maximally 11 years of age
* Diagnosis of asthma
* Baseline lung function tests as determined by protocol and required and received daily treatment with inhaled corticosteroids for at least 4 weeks prior to study start

Exclusion Criteria:

* Has required treatment with any non-inhaled corticosteroids within the previous 4 weeks, has sensitivity to drugs specified in the protocol or requires treatment with beta-blockers
* Has had cancer in the previous 5 years or has a significant disease that may put the patient at risk in this study

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 175 (Estimated)
Dates: Start 2002-07; Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Long term safety profile of Symbicort compared to Pulmicort as determined by safety assessments detailed in the protocol | 4 assessments within 26 week treatment period

SECONDARY OUTCOMES:
Compare health economic outcomes and quality of life between patients treated with Symbicort and Pulmicort | 4 assessments within 26 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Bonuccelli, Study Director — AstraZeneca